CLINICAL TRIAL: NCT02014090
Title: Acute Cardiovascular Effects of External Counterpulsation (ECP) in Comparison With Physical Exercise in Healthy Individuals
Brief Title: Acute Hemodynamic and Biological Effects of ECP and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Christian Seiler, Prof Dr med, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 177/07
Record Dates: First submitted 2011-04-05; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Patients With Stable Coronary Artery Disease
Keywords: ECP; Endurance exercise; myocardial perfusion
MeSH Terms: interventions — Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- half supine bicycle Exercise (Active Comparator): 60 minutes of half supine bicycle exercise with submaximal workload
  Interventions: Other: Hemodynamic and biological measurements
- ECP (Active Comparator): 90 minutes of ECP
  Interventions: Other: Hemodynamic and biological measurements

INTERVENTIONS:
Other: Hemodynamic and biological measurements — by MCE, PWA, Doppler, Multiplex, FACS

SUMMARY:
The purpose of this study in humans with stable coronary artery disease (CAD) treatable by percutaneous intervention (PCI) is to evaluate the efficacy of Enhanced External Counterpulsation (EECP) with regard to coronary collateral growth.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, written informed consent to participate in the study

Exclusion Criteria:

* 1. Pregnancy (serum β-HCG<2 IU/l for all female volunteers)

Baseline History:

1. Endurance exercise 5 days before and the days between the exams
2. History of cardiovascular disease or surgery, including arterial hypertension, Raynaud phenomenon, recurrent migraine, or any cardiac rhythm disorder
3. History of metabolic disorder, particularly diabetes mellitus
4. History of respiratory, renal, hepatic or cerebral disease
5. Allergic reactions to Luminity or its components
6. Cardiovascular medication
7. Illness characterized by acute phase response
8. Anaemia with haemoglobin levels < 110 g/L

Baseline Physical Examination:

1. Peripheral artery disease

Baseline Echocardiogram:

1. Valvular heart disease
2. Aortic aneurysm (any abnormality of ascending aorta, aortic arch or descending aorta)
3. Intra- or extracardiac shunt
4. Systolic or diastolic left ventricular (LV) dysfunction
5. LV-hypertrophy
6. Pulmonary arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Myocardial Blood Flow (MBF) measurement by Myocardial Contrast Echocardiography (MCE) | During ECP respectively Bicycle Exercise, expected to be on average 90 minutes

SECONDARY OUTCOMES:
Puls Wave Velocity Analysis | At baseline & post intervention, expected to be on average 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Gloekler, MD, Principal Investigator — University of Bern; Stefano de Marchi, MD, Principal Investigator — University of Bern; Stefano Rimoldi, MD, Principal Investigator — University of Bern; Christian Seiler, MD, Study Director — University of Bern
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland